CLINICAL TRIAL: NCT06474962
Title: Cardiorespiratory Fitness and Health Parameters in E-cigarrete Users: Impact of a Short Term Pause in Consumption
Acronym: EXERVAPE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Bruno Gualano, Associate Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 71092523.7.0000.0068
Record Dates: First submitted 2024-06-04; First posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Electronic Nicotine Delivery Systems
Keywords: vaping; e-cigarette
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pause (Experimental): Individuals will attempt to halt e-cigarette consumption for 7 days
  Interventions: Behavioral: Pause
- Control (No Intervention): Individuals will continue habits as usual

INTERVENTIONS:
Behavioral: Pause — 7 days of no e-cigarette consumption
  Arms: Pause

SUMMARY:
Goal: Investigate the health effects of electronic cigarettes (e-cigarettes) and whether a short break from using them can improve health.

Participants:

Up to 148 people (74 who use e-cigarettes and 74 who don't) Age and sex will be matched between the groups.

Study Design:

Two connected studies:

Observational Study: Compares general health (including lung function, heart health, blood pressure, and inflammation) of e-cigarette users to non-smokers.

Clinical Trial: E-cigarette users will be randomly assigned to either:

Take a 7-day break from e-cigarettes (intervention group) Continue using e-cigarettes as usual (control group) Both groups will have their health measured before and after the 7-day period. Main Outcome: How well your heart and lungs work during exercise.

Other Outcomes: Lung function, blood vessel function, risk factors for heart disease, and body measurements.

Why is this study important?

E-cigarettes are becoming more popular, but their health effects are unknown. This study will provide new information on whether e-cigarettes harm your health and if quitting for a short time can improve it.

This information can be used to create better public health policies about e-cigarettes.

DETAILED DESCRIPTION:
The emergence of electronic smoking devices is a recent and scientifically underexplored phenomenon. These devices were initially thought of as a harm-reduction strategy in cigarette smokers, a purpose for which there is still no definitive evidence of effectiveness. Preliminary but consistent findings in the literature suggest the possibility of detrimental health effects to e-cigarette users. Despite being prohibited for sale in the country, electronic cigarettes are easily accessible, in an unregulated manner. The increasing number of users, approaching one million according to recent data, and the uncertainties regarding the composition, manufacturing quality, and potential long-term effects of exposure to the vapor they produce, make the use of electronic cigarettes an emerging issue in Brazilian public health. Based on the aforementioned issues, exploring the potential effects of this new health-related behavior is urgent. Thus, the present proposal describes a research project envisioning the execution of two interconnected studies: (1) an observational cross-sectional analysis, in an exposed-control design, evaluating general health parameters of electronic cigarette users compared to non-smoking control individuals, matched by sex and age; and (2) an intervention study nested within the first study, designed as a randomized clinical trial, with electronic cigarette users assigned to a group that will take a 7-day pause from using these devices, compared to a control group that will not undergo any intervention. The studies were designed with cardiorespiratory fitness - measured by a maximum exercise cardiopulmonary test (ergospirometry) - as the primary outcome. The sample size calculated for the cross-sectional study comprises 148 individuals (74 per group), and the intended sample for the randomized clinical trial consists of the 74 electronic cigarette users already recruited for the cross-sectional study. The secondary outcomes of both studies are related to cardiorespiratory parameters, pulmonary function (spirometry), vascular function (endothelial function and tissue oxygenation), cardiovascular risk (lipid profile and blood pressure), inflammatory markers, and anthropometric measurements. The statistical analyses will be performed using Analysis of Covariance (ANCOVA), with physical activity level as a covariate for the cross-sectional study, and Generalized Estimating Equations (GEE), with initial oxygen consumption value as a covariate for the clinical trial. The investigators expect that the proposed studies yield new and relevant information regarding the potential harmful effects of electronic cigarettes, as well as the possibility of reversing these effects through refraining from their consumption. The novelty of the studies, the urgency of the topic, the boldness of the experimental approaches, and the high immediate applicability of the findings are highlighted in this proposal, with the potential to support public health policies concerning this relevant issue.

ELIGIBILITY:
Inclusion Criteria:

* 14 years of age or older
* Reporting using nicotine electronic cigarettes (e-cigarettes)
* Serum cotinine levels equal to or greater than 3 ng/mL

Exclusion Criteria:

* Contraindications for maximum exercise testing or any of study procedures
* Use of any smoking product except e-cigarette (combustible cigarette, cigar, hookah, marijuana, etc.)

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Maximal oxygen consumption | Baseline
  Maximal cardiorespiratory fitness assessed in a treadmill test
Maximal oxygen consumption | 7 days
  Maximal cardiorespiratory fitness assessed in a treadmill test

SECONDARY OUTCOMES:
Pulmonary function | Baseline
  Assessed through spirometry analysis of flow volume loops patterns
Pulmonary function | 7 days
  Assessed through spirometry analysis of flow volume loops patterns
Endothelial function | Baseline
  Assessed through ultrasonography of brachial artery
Endothelial function | 7 days
  Assessed through ultrasonography of brachial artery
Lipid profile | Baseline
  Blood concentrations of HDL cholesterol, LDL cholesterol, total cholesterol and tryglicerides
Lipid profile | 7 days
  Blood concentrations of HDL cholesterol, LDL cholesterol, total cholesterol and tryglicerides
Health-related quality of life | Baseline
  Assessed through "Short-form 36" questionnaire
Health-related quality of life | 7 days
  Assessed through "Short-form 36" questionnaire
Anxiety symptoms | Baseline
  Assessed through Beck's Anxiety Inventory
Anxiety symptoms | 7 days
  Assessed through Beck's Anxiety Inventory
Blood pressure | Baseline
  Office blood pressure measured with automated oscillometric device
Inflammatory status | Baseline
  Measured by blood concentration of inflammatory markers: interleukins 6 and 10, interferon-gamma, c-reactive protein and tumoral necrosis factor alpha
Inflammatory status | 7 days
  Measured by blood concentration of inflammatory markers: interleukins 6 and 10, interferon-gamma, c-reactive protein and tumoral necrosis factor alpha

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Gualano, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Clinical Hospital of the School of Medicine, University of Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared in accordance with institutional and legal requirements and will be provided upon reasonable request.
Time Frame: Data will be available upon the publication of first study report containing the study's primary outcome and will be kept available indefinitely.
Access Criteria: E-mail to study's principal investigator requesting data will be analyzed by the study team.